CLINICAL TRIAL: NCT02171780
Title: A Randomised, Double-blind, Placebo-controlled (Within Dose Groups) Study to Assess Safety, Tolerability and Pharmacokinetics of Single Rising Inhaled Doses (0.5 μg to 70 μg Administered With the Respimat®) of BI 1744 CL in Healthy Male and Female Volunteers
Brief Title: A Study to Assess Safety, Tolerability and Pharmacokinetics of Single Rising Inhaled Doses of BI 1744 CL in Healthy Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1222.1
Record Dates: First submitted 2014-06-20; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
MeSH Terms: interventions — olodaterol

ARMS (2):
- BI 1744 CL single rising doses (Experimental)
  Interventions: Drug: BI 1744 CL
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BI 1744 CL
  Arms: BI 1744 CL single rising doses
Drug: Placebo
  Arms: Placebo

SUMMARY:
To investigate safety, tolerability, and pharmacokinetics of BI 1744 CL

ELIGIBILITY:
Inclusion Criteria:

* The subject is healthy based upon a complete medical history, including the physical examination, regarding vital signs (BP, PR), 12-lead ECG measurement, and clinical laboratory tests. There is no finding deviating from normal and of clinical relevance. There is no evidence of a clinically relevant concomitant disease
* The subject is at least 21 years old and not older than 50 years
* The subject's body mass index (BMI) is at least 18.5 kg/m2 and less than 30 kg/m2
* The subject has signed and dated a written informed consent prior to admission to the study in accordance with GCP (Good Clinical Practice) and the local legislation

Exclusion Criteria:

* The subject has any finding of the medical examination (including BP, PR, and ECG measurements) deviating from normal and of clinical relevance
* The subject had a surgery of gastrointestinal tract (except appendectomy)
* The subject has a diagnosis of gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* The subject has a diagnosis of diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* The subject has a history of relevant orthostatic hypotension, fainting spells or blackouts
* The subject has a diagnosis of chronic or relevant acute infections
* The subject has a history of relevant allergy/hypersensitivity (including allergy to the drug or its excipients) as judged clinically relevant by the investigator
* The subject has taken drugs with a long half-life (>24 hours) within at least one month or less than 10 half-lives of the respective drug prior to randomisation
* The subject has used drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to randomisation
* The subject has participated in another trial with an investigational drug within two months prior to randomisation
* The subject is a heavily smoker (>10 cigarettes or >3 cigars or >3 pipes/day)
* The subject is not able to refrain from smoking on trial days as judged by the investigator
* The subject uses more than 60 g alcohol a day)
* The subject uses drugs
* The subject has donated more than 100 mL blood within four weeks prior to randomisation
* The subject has performed excessive physical activities within one week prior to randomisation
* The subject has a laboratory value outside the reference range that is of clinical relevance
* The subject is not able to comply with dietary regimen of the study centre.

The following exclusion criteria were specific for this study due to the known class side effect profile of ß2-mimetics:

* The subject has a diagnosis of asthma or history of pulmonary hyperreactivity
* The subject has a diagnosis of hyperthyrosis
* The subject has a diagnosis of allergic rhinitis in need of treatment
* The subject has a diagnosis of clinically relevant cardiac arrhythmia
* The subject has a diagnosis of paroxysmal tachycardia (>100 beats per minute).

For female subjects:

* Pregnancy
* Positive pregnancy test
* No adequate contraception e.g. oral contraception, sterilisation, IUD (intrauterine device). Females who are not surgically sterile will be asked to additionally use barrier contraception methods (e.g. condoms) prior to administration of study medication, during the study and at least one month after release from the study
* Inability to maintain this adequate contraception during the whole study period
* Lactation period

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 122 (Actual)
Dates: Start 2005-02; Primary Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Number of patients with abnormal findings in physical examination | 12 days after drug administration
Number of patients with clinically significant changes in vital signs | Baseline, up to 12 days after drug administration
Change in orthostasis test parameters | Baseline, up to 24 hours after drug administration
Number of patients with abnormal changes in laboratory parameters | Baseline, up to 12 days after drug administration
Change in oral body temperature | Baseline, up to 24 hours after drug administration
Number of patients with abnormal changes in 12-lead ECG (electrocardiogram) parameters | Baseline, up to 12 days after drug administration
Number of patients with adverse events | Up to 12 days
Change in tremormetry parameters | Baseline, up to 24 hours after drug administration
Number of patients with abnormal findings of oropharyngeal inspection | Baseline, up to 24 hours after drug administration
Number of patients with abnormal findings of pulmonary auscultation | Baseline, up to 24 hours after drug administration
Change in airway resistance (Raw), as measured by body plethysmography | Baseline, up to 24 hours after drug administration
Assessment of tolerability by investigator on a 4-point scale | 12 days after drug administration

SECONDARY OUTCOMES:
Area under the concentration-time curve of BI 1744 CL in plasma over the time interval from 0 to the time of the last quantifiable data point (AUC0-tz) | Up to 96 hours after drug administration
Area under the concentration-time curve of BI 1744 CL in plasma over the time interval from 0 to 24 hours (AUC0-24) | Up to 96 hours after drug administration
Maximum concentration of BI 1744 CL in plasma (Cmax) | Up to 96 hours after drug administration
Time from dosing to maximum concentration (tmax) | Up to 96 hours after drug administration
Amount of BI 1744 CLeliminated in urine from the time point t1 to time point t2 (Aet1-t2) | Up to 96 hours after drug administration
Fraction of BI 1744 CL eliminated in urine from time point t1 to time point t2 (fet1-t2) | Up to 96 hours after drug administration
Renal clearance of BI 1744 CL from 0 to 24 hours (CLR,0-24) | Up to 24 hours after drug administration
Terminal rate constant of BI 1744 CL in plasma (λz) | Up to 96 hours after drug administration
Terminal half-life of BI 1744 CL in plasma (t½) | Up to 96 hours after drug administration
Area under the concentration-time curve of BI 1744 CL in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) | Up to 96 hours after drug administration
AUC0-tz over AUC0-∞ (%AUC0-tz) | Up to 96 hours after drug administration
Mean residence time of BI 1744 CL in the body after inhalation (MRTih) | Up to 96 hours after drug administration
Apparent clearance of BI 1744 CL in the plasma after extravascular administration (CL/F) | Up to 96 hours after drug administration
Apparent volume of distribution of BI 1744 CL during the terminal phase λz following an extravascular dose (Vz/F) | Up to 96 hours after drug administration